CLINICAL TRIAL: NCT05394623
Title: Prevalence and Burden of Hepatitis D Virus Infection in China Through Preoperative Examination Test (Predict Study)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-8764
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Hepatitis D; Hepatitis B; Antibodies; Anti-D; RNA Virus Infections
MeSH Terms: conditions — Hepatitis D; Hepatitis B; RNA Virus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HDV-Ab (IgG), HDV-RNA, RNA genotype — Anti-HDV was evaluated semiquantitatively by means of end-point dilutions. Quantitative HDV-RNA was performed by means of LightCycler 2.0. Genotyping of HDV was performed by direct sequencing of the delta antigen region.

SUMMARY:
In China, there is no recommendation for Hepatitis D virus (HDV) screening, but the fact is estimated that one-third of the world's population of individuals with chronic Hepatitis B virus (HBV) infection live in China while we do not know the prevalence of co-infection of HBV/HDV in China. So far, no nationwide study has been undertaken to evaluate the epidemiology of hepatitis D, on the other hand, reports of HDV infection rate in different regions of China are not consistent because of the different detection methods and detection objects. Here, we plan to test HDV-Ab/RNA for 5000 HBsAg reactive samples from 10 major tertiary hospital and to know the prevalence and disease burden of HDV in China.

ELIGIBILITY:
Inclusion Criteria:

1. Positive HBV surface antigen (HBsAg)
2. Age 18 yeas and above

Exclusion Criteria:

1. Severe cardiac, renal, respiratory, hematological, or psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatitis D virus-infected patients in HBsAg positive population from 10 hospitals located in 5 diſferent geographical areas (North, South, East, West and Central) in China.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
HDV seroprevalence and HDV RNA prevalence amongst HBsAg positive carriers in China. | 3 months
  Briefly, serum samples were tested undiluted, and after dilution of 1:10, 1:100, 1:1,000, 1:5,000, 1:10,000, 1:50,000, and was considered the highest dilution with a S/Co value >1.0. The detection system consisted of a competitive enzyme immunoassay, in which Anti-HDV antibodies (IgG/IgM), if present in the sample, compete with a virus-specific human polyclonal IgG, labeled with peroxidase (HRP), for a ţxed amount of full-length rec-HDV coated on the microplate. Qualitative HDV RNA was determined by in-house Polymerase Chain Reaction (PCR). Quantitative HDV-RNA was performed by means of LightCycler 2.0 (lower limit of detection 10 copies/reaction).

SECONDARY OUTCOMES:
The distribution of HDV genotypes in China | 3 months
  Genotyping of HDV was performed by direct sequencing of the delta antigen region.